CLINICAL TRIAL: NCT01457014
Title: BiPAP Adaptive Servo-Ventilation (AutoSV) Therapy in Patients With Chronic Pain and Sleep Disordered Breathing (SDB)
Brief Title: Sleep Disordered Breathing and Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SDBPM-2011-01
Record Dates: First submitted 2011-09-30; First posted 2011-10-21 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-01

CONDITIONS: Sleep Apnea Syndromes
Keywords: chronic pain; sleep disordered breathing; Opioids
MeSH Terms: conditions — Sleep Apnea Syndromes; Chronic Pain | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- servo ventilation auto mode (Active Comparator): Inspiratory and expiratory pressures automatically determined by the servo ventilation device.
  Interventions: Device: servo ventilation auto; Device: Continuous positive airway pressure; Device: servo ventilation manual
- Continuous positive airway pressure (Active Comparator): Airway pressure delivered at a constant pressure level.
  Interventions: Device: Continuous positive airway pressure; Device: servo ventilation manual
- servo ventilation manual (Active Comparator): Inspiratory and expiratory pressures automatically determined by the servo ventilation device with mandatory minimal inspiratory minus expiratory pressure difference.
  Interventions: Device: servo ventilation manual

INTERVENTIONS:
Device: servo ventilation auto — Expiratory pressure automatically adjusted to stabilize the upper airway. Inspiratory pressure automatically adjusted to deliver consistent peak flow.
  Arms: servo ventilation auto mode
Device: Continuous positive airway pressure — continuous positive airway pressure
  Other Names: CPAP
  Arms: Continuous positive airway pressure; servo ventilation auto mode
Device: servo ventilation manual — servo ventilation titrated in manual mode

SUMMARY:
The purpose of this study is to evaluate positive pressure in patients with chronic pain taking opioid medications who have sleep disordered breathing.

DETAILED DESCRIPTION:
Purpose: Opioid treatment of non-malignant chronic pain can result in hypoxemia, hypercarbia, and central sleep apnea. The aim of this study was to determine the initial efficacy of auto servo-ventilation (ASV) and after 3 months of home use.

Methods: This prospective multicenter interventional study recruited chronic pain patients prescribed ≥100 morphine equivalents for at least 4 months.

Participants: Following full-night polysomnography (PSG) to confirm the presence of sleep-disordered breathing, patients were randomized to three additional full-night-attended PSGs with continuous positive airway pressure (CPAP), ASV, and servo-ventilation with an initial mandatory pressure support of 6 cm water (H2O) ASV manual Minimum Pressure Support (PSmin). Following the PSGs, patients were sent home with EncoreAnywhere and ASV with or without mandatory pressure support.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, ages 21-70.
2. Able to provide written informed consent.
3. Diagnosis of chronic non-malignant pain (pain present for ≥ 6 months).
4. Stable regimen of opioids (oral, transdermal, and/or intravenous) for chronic pain for at least 4 weeks prior to study participation with a prescribed opioid dose equal to at least 100 milliequivalents of morphine per 24 hours (Appendix 1).
5. Agreement to undergo an in-lab Diagnostic polysomnography (PSG) demonstrating an Apnea-Hypopnea Index (AHI) of at least 20 and Central Apnea Index (CAI) ≥ 10 events per hour of sleep OR at least 25% of Total Sleep Time (TST) below 90% Oxygen Saturation (SAO2) saturation and AHI ≥ 10
6. Agreement to undergo 3 full-night, in-lab PSG's on positive airway pressure therapy.
7. Agreement to undergo breathalyzer testing prior to each PSG visit
8. Ability to provide reliable documentation of opioid medications (ex. Pharmacy records) as treatment for chronic pain for the previous 30 days.
9. Willingness to undergo urine drug screening.

Exclusion Criteria:

1. Participation in other interventional, sleep or pharmaceutical related research studies within 30 days prior to giving consent.
2. Workers with variable shift schedules.
3. Previous treatment with positive airway pressure therapy within 90 days of providing consent.
4. Participants with any conditions in which positive airway pressure is medically contraindicated (e.g. recent pneumothorax, systolic BP < 80 mmHg).
5. BMI > 40
6. Unwilling to wear PAP.
7. Any surgery involving the upper airway, eye, nose, sinuses or middle ear within the last 90 days.
8. Major or poorly managed medical or psychiatric condition that would interfere with the demands of the study, to the use of positive airway pressure, or the ability to complete the study.
9. Previous diagnosis of severe chronic obstructive pulmonary disease (COPD) with an forced expiratory volume at one second (FEV1) < 1 liter or less than 50% predicted
10. Presence of elevated arterial carbon dioxide levels while awake (PaCO2 ≥ 50mmHg) due to intrinsic lung disease, neuromuscular or musculoskeletal disorders.
11. Participants currently prescribed 24 hour oxygen therapy (nocturnal O2 therapy for obstructive sleep apnea (OSA) treatment is allowed)
12. Females who are pregnant or, if of child bearing potential, not currently using medically reliable birth control methods.
13. Participants prescribed opioids for reasons other than the management of chronic, non-malignant pain.
14. Failure of two consecutive breathalyzer tests from study PSG nights
15. Periodic Limb Movements (PLM's) with arousals > 15

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wylie, MD, Principal Investigator — Arkansas Center of Sleep Medicine; Vernon Pegram, PhD, Principal Investigator — Sleep D/O Center of Alabama; Mark Muehlbach, PhD, Principal Investigator — Clayton Sleep Institute; Russell Rosenberg, MD, Principal Investigator — NeuroTrials Research, Inc.
Locations (4):
- United States (4):
  - Sleep D/O Center of Alabama, Birmingham, Alabama
  - Arkansas Center for Sleep Medicine, Little Rock, Arkansas
  - NeuroTrials Research Inc., Atlanta, Georgia
  - Clayton Sleep Institute, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from pain treatment centers and clinics by either Pain Center/Clinic staff or staff from a Sleep Testing facility.
Pre-assignment Details: 74 participants were screened; 40 were excluded after completing the diagnostic PSG (did not meet the inclusion/exclusion criteria).
Groups:
- Diagnostic Polysomnography (PSG): A Diagnostic PSG was performed using the core equipment available to determine eligibility into the overnight portion of the study.
- Continuous Positive Airway Pressure (CPAP): Airway pressure delivered at a constant pressure level.
  CPAP: continuous positive airway pressure
  servo ventilation manual: servo ventilation titrated in manual mode
- Servo Ventilation Auto Mode (autoSV): Inspiratory and expiratory pressures automatically determined by the servo ventilation device.
  servo ventilation auto: Expiratory pressure automatically adjusted to stabilize the upper airway. Inspiratory pressure automatically adjusted to deliver consistent peak flow.
  CPAP: continuous positive airway pressure
  servo ventilation manual: servo ventilation titrated in manual mode
- Servo Ventilation Manual (Manual SV): Inspiratory and expiratory pressures automatically determined by the servo ventilation device with mandatory minimal inspiratory minus expiratory pressure difference.
  servo ventilation manual: servo ventilation titrated in manual mode
Period: First Night
Arm/Group | Diagnostic Polysomnography (PSG) | Continuous Positive Airway Pressure (CPAP) | Servo Ventilation Auto Mode (autoSV) | Servo Ventilation Manual (Manual SV)
Started | 74 | 0 | 0 | 0
Completed | 34 | 0 | 0 | 0
Not Completed | 40 | 0 | 0 | 0
Not completed — Didn't meet inclusion/exclusion criteria | 37 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0
Period: Second Night
Arm/Group | Diagnostic Polysomnography (PSG) | Continuous Positive Airway Pressure (CPAP) | Servo Ventilation Auto Mode (autoSV) | Servo Ventilation Manual (Manual SV)
Started | 0 (The Diagnostic PSG was only completed on the First night) | 12 (Participants were randomized to different arms for each overnight stay: CPAP, Auto SV, Manual SV.) | 11 (Participants were randomized to different arms for each overnight stay: CPAP, Auto SV, Manual SV.) | 11 (Participants were randomized to different arms for each overnight stay: CPAP, Auto SV, Manual SV.)
Completed | 0 (The Diagnostic PSG was only completed on the First night) | 12 | 11 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Third Night
Arm/Group | Diagnostic Polysomnography (PSG) | Continuous Positive Airway Pressure (CPAP) | Servo Ventilation Auto Mode (autoSV) | Servo Ventilation Manual (Manual SV)
Started | 0 (The Diagnostic PSG was only completed on the First night) | 11 (Participants were randomized to different arms for each overnight stay: CPAP, Auto SV, Manual SV.) | 11 (Participants were randomized to different arms for each overnight stay: CPAP, Auto SV, Manual SV.) | 12 (Participants were randomized to different arms for each overnight stay: CPAP, Auto SV, Manual SV.)
Completed | 0 (The Diagnostic PSG was only completed on the First night) | 11 | 11 | 12
Not Completed | 0 | 0 | 0 | 0
Period: Fourth Night
Arm/Group | Diagnostic Polysomnography (PSG) | Continuous Positive Airway Pressure (CPAP) | Servo Ventilation Auto Mode (autoSV) | Servo Ventilation Manual (Manual SV)
Started | 0 (The Diagnostic PSG was only completed on the First night) | 11 (Participants were randomized to different arms for each overnight stay: CPAP, Auto SV, Manual SV.) | 12 (Participants were randomized to different arms for each overnight stay: CPAP, Auto SV, Manual SV.) | 11 (Participants were randomized to different arms for each overnight stay: CPAP, Auto SV, Manual SV.)
Completed | 0 (The Diagnostic PSG was only completed on the First night) | 11 | 12 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of participants that completed the baseline PSG and were randomized for the study.
Groups:
- Total Group: 34 subjects completed part 1 of the study which consisted of diagnostic PSG screening and met all inclusion/exclusion criteria
Arm/Group | Total Group
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 15
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 31
  African American | 3
Region of Enrollment [Number; unit: participants]
  United States | 34
Morphine equivalents [Mean (Standard Deviation); unit: mEq] — 1. Calculate the total daily dose (24h) for each long acting and short acting opioid.
  2. Divide the total daily dose for each opioid by its equianalgesic dose (ED) (see chart) to get the equianalgesic dose units (EDU).
  3. Add the EDU for each opioid to get the total EDU for all opioids.
  4. Multiply the total EDU by 30 mg to get the morphine equivalent dose (meq of morphine).
  Opioid- ED Morphine- 30 Hydrocodone- 30 Oxycodone- 20 Hydromorphone- 7.5 Codeine- 200 Methadone- 2-4 (chronic opioid users) Meperidine- 300 Tramadol- 1:5 ratio whereas10 mg morphine = 50mg Tramadol
  mEq | 390.1 (338.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Sleep Related Events Per Hour
Description: The number of Apnea-Hypopnea Events, Central Apneas, Obstructive Apneas and Hypopneas were compared among no treatment, CPAP, Auto SV and Manual SV.
Time Frame: four full night Polysomnography (PSG's)
Population: After the Diagnostic Polysomnography (PSG) each participant completed a night in each arm.
Measure: Mean (Standard Deviation); unit: events/hour
Groups:
- Diagnostic Polysomnography (PSG): Baseline overnight Polysomnography (PSG)
- CPAP: Airway pressure delivered at a constant pressure level.
  CPAP: continuous positive airway pressure
  servo ventilation manual: servo ventilation titrated in manual mode
- Servo Ventilation Auto Mode: Inspiratory and expiratory pressures automatically determined by the servo ventilation device.
  servo ventilation auto: Expiratory pressure automatically adjusted to stabilize the upper airway. Inspiratory pressure automatically adjusted to deliver consistent peak flow.
  CPAP: continuous positive airway pressure
  servo ventilation manual: servo ventilation titrated in manual mode
Arm/Group | Diagnostic Polysomnography (PSG) | CPAP | Servo Ventilation Auto Mode | Servo Ventilation Manual
Number analyzed (Participants) | 31 | 31 | 31 | 31
events/hour
  Apnea-hyopnea index | 38.8 (31.1) | 17.4 (20.1) | 4.5 (7.3) | 7.6 (16.7)
  Central Apnea Index | 16.1 (18.8) | 8.4 (12.4) | 0.2 (0.8) | 0.2 (0.9)
  Obstructive Apnea Index | 9.7 (6.3) | 4.5 (6.3) | 0.3 (0.5) | 0.5 (1.1)
  Hypopnea Index | 14.8 (12.6) | 4.5 (5.1) | 4.6 (7.4) | 7.9 (16.2)
Statistical Analysis 1: Comparison: CPAP vs Servo Ventilation Auto Mode vs Servo Ventilation Manual; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); p values have undergone Bonferroni adjustment for Central Apnea Index (CAI), Obstructive Apnea Index (OAI) and Hypopnea Index (HI)

2. Secondary Outcome: Percent Oxygen Saturation
Description: Oxygen Saturation were compared among using no treatment, CPAP, Auto SV and Manual SV.
Time Frame: four full night Polysomnography (PSG's)
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Groups:
- Diagnostic PSG: Baseline overnight PSG.
Arm/Group | Diagnostic PSG | CPAP | Servo Ventilation Auto Mode | Servo Ventilation Manual
Number analyzed (Participants) | 31 | 31 | 31 | 31
percentage of oxygen saturation
  Av. O2 saturation | 92.9 (3.4) | 94.6 (2.3) | 94.6 (2.6) | 94.5 (3.2)
  Min. O2 saturation | 79.9 (7.8) | 85.5 (6.0) | 82.9 (16.2) | 79.7 (22.8)
Statistical Analysis 1: Comparison: CPAP vs Servo Ventilation Auto Mode vs Servo Ventilation Manual; Test type: Superiority or Other; p = 0.627, Wilcoxon (Mann-Whitney) — p value has undergone Bonferroni adjustment. P-Value applies to Av. 02 saturation; p value has undergone Bonferroni adjustment

3. Secondary Outcome: Number of Arterial Oxygen Saturation Per Hour
Description: Arterial Oxygen Saturation was compared among using no treatment, CPAP, Auto SV and Manual SV.
Time Frame: four full night Polysomnography (PSG's)
Measure: Mean (Standard Deviation); unit: times per hour
Arm/Group | Diagnostic PSG | CPAP | Servo Ventilation Auto Mode | Servo Ventilation Manual
Number analyzed (Participants) | 31 | 31 | 31 | 31
times per hour | 32.8 (29.2) | 15.1 (20.2) | 5.9 (8.6) | 9.5 (19.2)
Statistical Analysis 1: Comparison: CPAP vs Servo Ventilation Auto Mode vs Servo Ventilation Manual; Test type: Superiority or Other; p = .161, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Total Group
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 14/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total Group (N=34)
Common Cold (Immune system disorders) | 3
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Sinus Infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 4
Ear Infection (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No